CLINICAL TRIAL: NCT03129386
Title: Defining the Normal Range for Maximal Sniff Diaphragm Thickening Fraction
Acronym: SNIFF II
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Ewan Goligher, Intensivist, University Health Network, Toronto
Other Study IDs: 15-8998-AE
Record Dates: First submitted 2017-04-04; First posted 2017-04-26 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Diaphragm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is investigating the normal range of maximal diaphragm thickness during a sniff inspiratory manoeuvre using ultrasound in healthy subjects stratified by age and gender.

DETAILED DESCRIPTION:
Diaphragm dysfunction is associated with poor clinical outcomes in critically ill patients but is difficult to diagnose. Traditionally, diaphragm function is measured by evaluating inspiratory muscle strength via maximal inspiratory pressure (MIP). However, this technique relies on a volitional maximal effort and can be challenging for patients to perform.

An alternative to measuring inspiratory muscle strength is the sniff inspiratory pressure approach. During short, sharp sniffs, the diaphragm is maximally activated.

Currently, there are no reported values of the normal range of maximal diaphragm thickness during a sniff maneuver. This study will define the normal range of values for sniff maximal diaphragm thickening fraction, maximal thickening against an occluded airway, and diaphragm thickening during resting tidal breathing in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age

Exclusion Criteria:

* Antecedent history of neuromuscular or cardiorespiratory disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adult subjects with no antecedent history of neuromuscular or cardiorespiratory disease.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-06-08 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Sniff diaphragm thickening fraction | Day 1
  Thickening of the diaphragm during an inspiratory sniff
Maximal diaphragm thickening fraction | Day 1
  Thickening of the diaphragm during a maximal inspiratory effort
Resting tidal thickening fraction | Day 1
  Thickening of the diaphragm during resting tidal breathing

CONTACTS AND LOCATIONS:
Overall Officials: Ewan C Goligher, MD, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Currently, there is no plan to make data IPD available to others.